CLINICAL TRIAL: NCT00127608
Title: An Open, Prospective, Non-prophylactic, Non Therapeutic Study for the Detection and Characterisation of Varicella Zoster Virus Collected From Dermal Lesions of Patients Who Are Diagnosed of Having Varicella/Breakthrough Varicella
Brief Title: Detection and Characterisation of Varicella Zoster Virus From Dermal Lesions of Chickenpox-infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 103815
Record Dates: First submitted 2005-08-04; First posted 2005-08-08 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2018-08

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox

ARMS (1):
- Varicella Group (Experimental): Subjects aged between 0 and 16 years of age, with clinically-diagnosed primary varicella disease.
  Interventions: Procedure: Collection of clinical samples

INTERVENTIONS:
Procedure: Collection of clinical samples — The following samples were obtained from each subject:
  * Vesicle fluid (VF) and vesicle swabs (VS) from four vesicles (for a total of eight samples)
  * Papule swabs (PS) from four papules
  * Crusts from two lesions
  * One throat swab (TS) Up to 15 samples were to be obtained for each subject, when possible. VFs, VSs, PSs, and crusts were either stored dry or in liquid medium. TS samples were stored in liquid medium.
  After extraction of DNA, samples were tested for the presence of varicella virus using a Quantitative Polymerase Chain Reaction (Q-PCR) technique.

SUMMARY:
This study is conducted in order to collect clinical samples from patients who are diagnosed of having chickenpox infection. The results of this study will provide basic scientific information about chickenpox disease.

DETAILED DESCRIPTION:
The study involves NO therapeutic or prophylactic treatment nor further observation of the patients. There is no product to be tested in this study.

ELIGIBILITY:
Pediatric patients who are diagnosed of having varicella and are presenting varicella dermal lesions.

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2005-06-07 (Actual); Primary Completion 2006-07-13 (Actual); Study Completion 2006-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Similar numbers of subjects presenting with different varicella rash intensities were enrolled:
  * Severe: more than 150 lesions on multiple parts of the body; rash is mostly vesicular
  * Moderate: 51 to 150 lesions; rash is vesicular and/or maculopapular
  * Mild: 1-50 lesions; rash is maculopapular rather than vesicular
Pre-assignment Details: Out of 503 samples collected, 6 were not received from the investigator and 12 were insufficient samples. Hence only 485 samples were tested by Q-PCR.
  All 13 samples from 1 subject were VZV DNA negative, suggesting the subject did not have varicella. Therefore, this subject was not included in the final analyses and hence not completed.
Units Other Than Participants: samples
Period: Overall Study
Arm/Group | Varicella Group
Started | 36; 503 samples
Completed | 35; 472 samples
Not Completed | 1; 31 samples
Not completed — VZV DNA negative | 1

BASELINE CHARACTERISTICS:
Arm/Group | Varicella Group
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: Years] | 5.33 [0 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Viral Load: Number of Varicella Zoster Virus (VZV) Deoxyribonucleic Acid (DNA) Copies Per Clinical Sample
Description: The estimated means of the viral load in log10 values for each storage condition (dry and liquid) and each type of sample are presented with 95% confidence intervals
Time Frame: At Visit 1 (Day 0)
Population: One subject who was Varicella Zoster Virus (VZV) deoxyribonucleic acid (DNA)-negative in all samples taken, was considered not to have varicella and was not included in the analyses.
Measure: Log Mean (95% Confidence Interval); unit: VZV genome copies per sample
Units Other Than Participants: samples
Arm/Group | Varicella Group
Number analyzed (Participants) | 35
Number analyzed (samples) | 472
VZV genome copies per sample
  Vesicle fluid (dry storage): number analyzed (samples) | 65
  Vesicle fluid (dry storage) | 6.49 [4.58 to 7.58]
  Vesicle swab (dry storage): number analyzed (samples) | 63
  Vesicle swab (dry storage) | 6.46 [4.64 to 7.69]
  Papule swab (dry storage): number analyzed (samples) | 65
  Papule swab (dry storage) | 6.07 [3.93 to 7.43]
  Crust (dry storage): number analyzed (samples) | 22
  Crust (dry storage) | 6.02 [4.21 to 7.47]
  Vesicle fluid (liquid storage): number analyzed (samples) | 65
  Vesicle fluid (liquid storage) | 6.98 [5.74 to 7.91]
  Vesicle swab (liquid storage): number analyzed (samples) | 60
  Vesicle swab (liquid storage) | 6.98 [5.62 to 7.99]
  Papule swab (liquid storage): number analyzed (samples) | 68
  Papule swab (liquid storage) | 6.09 [5.03 to 8.21]
  Crust (liquid storage): number analyzed (samples) | 29
  Crust (liquid storage) | 7.08 [4.98 to 8.10]
  Throat swab (liquid storage): number analyzed (samples) | 35
  Throat swab (liquid storage) | 4.78 [2.93 to 7.15]

2. Primary Outcome: Viral Load: Number of Varicella Zoster Virus (VZV) Deoxyribonucleic Acid (DNA) Copies Per Clinical Sample by Storage Condition (Dry, Liquid)
Description: The estimated viral load was calculated by quantitative polymerase chain reaction assay (Q-PCR) in log10, as a mean number of viral copies per sample by storage conditions (dry, liquid). As throat swabs were not stored dry and the number of crust samples was lower than that of papules and vesicles, this analysis was done only on data from vesicle fluid, vesicle swabs and papule swabs.
Time Frame: At Visit 1 (Day 0)
Population: Only VZV DNA-positive samples were considered in this analysis.
Measure: Log Mean (95% Confidence Interval); unit: VZV genome copies per sample
Units Other Than Participants: samples
Arm/Group | Varicella Group
Number analyzed (Participants) | 35
Number analyzed (samples) | 383
VZV genome copies per sample
  Dry storage: number analyzed (samples) | 193
  Dry storage | 6.34 [6.18 to 6.50]
  Liquid storage: number analyzed (samples) | 190
  Liquid storage | 6.82 [6.67 to 6.98]
Statistical Analysis 1: Comparison: Varicella Group; Test type: Non-Inferiority — The mean viral load between samples stored in liquid and samples stored dry was compared; p < 0.0001, ANOVA; Tukey adjustments were made for all 2 by 2 comparisons; Geometric Mean Ratio = 0.33 — The Geometric Mean Ratio of the viral load was calculated for dry over liquid storage condition

3. Primary Outcome: Estimated Mean Viral Load (in log10) by Sample Types (Papule Swab, Vesicle Fluid and Vesicle Swab)
Description: The estimated viral load was calculated by quantitative polymerase chain reaction assay (Q-PCR) in log10, as a mean number of viral copies per sample by sample types (papule swab, vesicle fluid and vesicle swab).
  As throat swabs were not stored dry and the number of crust samples was lower than that of papules and vesicles, this analysis was done only on data from vesicle fluid, vesicle swabs and papule swabs.
Time Frame: At Visit 1 (Day 0)
Population: Only VZV DNA-positive samples were considered in this analysis.
Measure: Log Mean (95% Confidence Interval); unit: VZV genome copies per sample
Units Other Than Participants: samples
Arm/Group | Varicella Group
Number analyzed (Participants) | 35
Number analyzed (samples) | 383
VZV genome copies per sample
  Papule swab (Dry or Liquid storage): number analyzed (samples) | 130
  Papule swab (Dry or Liquid storage) | 6.29 [6.10 to 6.48]
  Vesicle fluid (Dry or Liquid storage): number analyzed (samples) | 130
  Vesicle fluid (Dry or Liquid storage) | 6.74 [6.54 to 6.92]
  Vesicle swab (Dry or Liquid storage): number analyzed (samples) | 123
  Vesicle swab (Dry or Liquid storage) | 6.72 [6.52 to 6.92]
Statistical Analysis 1: Comparison: Varicella Group; Test type: Non-Inferiority or Equivalence — Difference in mean viral load (in log10) (Papule swab minus Vesicle fluid); p = 0.0038, ANOVA; Tukey adjustments were made for the comparison; Mean Difference (Final Values) = -0.4451, 95% CI [-0.7690 to -0.1213]
Statistical Analysis 2: Comparison: Varicella Group; Test type: Non-Inferiority or Equivalence — Difference in mean viral load (in log10) (Papule swab minus Vesicle swab); p = 0.0060, ANOVA; Tukey adjustments were made for the comparison; Median Difference (Final Values) = -0.4320, 95% CI 2-sided [-0.7605 to -0.1035]
Statistical Analysis 3: Comparison: Varicella Group; Test type: Non-Inferiority or Equivalence — Difference in mean viral load (in log10) (Vesicle fluid minus Vesicle swab); p = 0.9952, ANOVA; Tukey adjustments were made for the comparison; Mean Difference (Final Values) = 0.00132, 95% CI 2-sided [-0.3171 to 0.3435]
Statistical Analysis 4: Comparison: Varicella Group; Geometric mean ratio of viral load (Papule swab over Vesicle fluid); Test type: Non-Inferiority or Equivalence — Geometric mean ratio of viral load (Papule swab over Vesicle fluid); ANOVA; Geometric mean ratio = 0.36, 95% CI 2-sided [0.17 to 0.76]
Statistical Analysis 5: Comparison: Varicella Group; Geometric mean ratio of viral load (Papule swab over Vesicle swab); Test type: Non-Inferiority or Equivalence — Geometric mean ratio of viral load (Papule swab over Vesicle swab); ANOVA; Geometric mean Ratio = 0.37, 95% CI 2-sided [0.17 to 0.79]
Statistical Analysis 6: Comparison: Varicella Group; Geometric mean ratio of viral load (Vesicle fluid over Vesicle swab); Test type: Non-Inferiority or Equivalence — Geometric mean ratio of viral load (Vesicle fluid over Vesicle swab); ANOVA; Geometric mean Ratio = 1.00, 95% CI 2-sided [0.48 to 2.21]

ADVERSE EVENTS:
Description: No solicited, unsolicited or serious adverse events were collected during this study.
Arm/Group | Varicella Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.